CLINICAL TRIAL: NCT00006440
Title: Feasibility Study of a Behavioral Intervention for Women at Persistent High Risk for HIV Infection
Brief Title: A Test of Behavioral Intervention for Women at High Risk for HIV Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: HIVNET 029
Record Dates: First submitted 2000-11-03; First posted 2001-08-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Risk Factors; Behavior Therapy; Substance-Related Disorders; Feasibility Studies
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders

SUMMARY:
The purpose of this study is to find out if it is possible to conduct a group counseling program for women at risk for HIV infection.

Women have been the fastest-growing group with new AIDS diagnoses. The need for ways to reduce HIV infection in women is urgent. It is important to reduce the risk of HIV infection through sexual contact, but it is also important to address drug use. Group counseling may be an effective method.

DETAILED DESCRIPTION:
Women have constituted the fastest-growing group of persons with new AIDS diagnoses for several years. The need to develop and evaluate interventions to reduce the incidence of HIV infection among women is urgent. The behavioral intervention method tested in this study integrates elements from diverse theories and empirical evidence for women to feel empowered to use methods of protection against disease. Although the overall objective of the study intervention is to reduce the risk of HIV infection through sexual contact, the intervention must also address drug usage among women.

Women are randomized in a 1 to 1 ratio to either the intervention or control condition. The Intervention Group participates in 4 group sessions over the course of 1 month and then in an additional reunion session approximately 1 month after the 4th group session. Sessions are 2.5 hours long and include 6 to 10 participants. The sessions involve talking about HIV, ways to avoid HIV, and ways women can support each other. All participants complete a short-term assessment visit 1 week after the 4th group intervention session. The Control Group does not participate in group sessions. All participants are paid for their time and effort.

ELIGIBILITY:
Inclusion Criteria

Women may be eligible for this study if they:

* Are at least 18 years old.
* Took part in the VPS2 study and completed 12 months of follow-up, or each participant must meet at least 1 of the following conditions: 1) has sex with an HIV-infected male; 2) has sex with a male who has injected drugs in the last 5 years; 3) has had sex with 5 or more male partners in the last year; 4) exchanged sex for money or drugs in the last year; 5) was diagnosed with syphilis, chlamydia, gonorrhea, first episode herpes, pelvic inflammatory disease, and/or trichomonas in the last year; or 6) used crack cocaine in the last year.
* Can speak English.
* Can give information for the purpose of locating.
* Have had at least 30 percent of vaginal or anal intercourse unprotected by condoms in the 6 months before the study.
* Are HIV-negative.

Exclusion Criteria

Women will not be eligible for this study if they:

* Have had sex with only 1 man for 2 years or more who is HIV-negative and does not inject drugs. The man should not have had sex with anyone else during this time.
* Have a mental condition that would interfere with the study.
* Have any other condition that would interfere with the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2000-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Gollub, Study Chair
Locations (1):
- Anne Colletti, Cambridge, Massachusetts, United States